CLINICAL TRIAL: NCT03496597
Title: Early Stage Retinal Abnormalities in Type 1 Diabetes, Screened With OCT Angiography.
Acronym: AwARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VERGES 2017
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: type 1 diabetes patients
  Interventions: Procedure: Retinal imaging assessment; Procedure: blood glucose holter
- Healthy controls: non diabetic control subjects of the same age
  Interventions: Procedure: Retinal imaging assessment
- Dyslipidemic controls: non-diabetic control participants with familial dyslipidemia
  Interventions: Procedure: Retinal imaging assessment

INTERVENTIONS:
Procedure: Retinal imaging assessment — * OCT-angiography
  * Automated measurement program: size of the avascular zone and perifoveolar vascular density of the superficial capillary plexus
  * Eye fundus photography: macular image
  * Measurement of the fractal dimension of the retinal foveolar retina from photographs of the fundus
Procedure: blood glucose holter — for 40 subjects, implantation of a blood glucose holter monitor for 7 days
  Groups: Patients

SUMMARY:
The improvement of imaging techniques in ophthalmology has made it possible to carry out a precise non-invasive study of the retinal microvascular network and to detect early abnormalities in retinal disorders. The presence of such early retinal abnormalities remains poorly known during type 1 diabetes and may be detected with OCT-angiography. Furthermore, the association with glycemic variability, likely to have deleterious effects on microvessels, has never been studied.

ELIGIBILITY:
Inclusion Criteria:

For the patient group

* Patient who has given consent

  * Type 1 diabetic patient, no retinopathy For the healthy control group
* Patient who has given consent
* Non-diabetic patient

For dyslipidemic control group:

* Person who has given consent
* Person with familial dyslipidemia

Exclusion Criteria:

For the patient group

* Presence of diabetic retinopathy
* Protected patient:

  * Minor patient
  * Pregnant, parturient or breastfeeding woman
  * Patient under legal protection (guardianship, curatorship, court decision)
  * Patient unable to express consent Person not affiliated to a health insurance scheme

For the healthy control group

* Ophthalmological history (vascular and degenerative macular conditions)
* Protected patient:

  * Minor patient
  * Pregnant, parturient or breastfeeding woman
  * Patient under legal protection (guardianship, curatorship, court decision)
  * Patient unable to express consent Person not affiliated to a social security scheme

For dyslipidemic control group:

* Ophthalmological history (vascular and degenerative macular conditions)
* Protected patient:

  * Minor patient
  * Pregnant, parturient or breastfeeding woman
  * Patient under legal protection (guardianship, curatorship, court decision)
  * Patient unable to express consent Person not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetes Type 1 patients followed in the Endocrinology Department of the CHU Dijon Bourgogne or in a diabetology surgery, and non-diabetic controls will be recruited in the Ophthalmology Department of the CHU Dijon Bourgogne
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
surface of the central retinal avascular zone | inclusion
  measurement of superficial capillary plexus

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France